CLINICAL TRIAL: NCT04150107
Title: A Phase 2 Randomized, Open Label Crossover Study to Compare ORMD-0801 Given Once Daily at Bedtime to ORMD-0801 Given Three Times Daily (45-90 Minutes Before Meals) in Subjects With Type 1 Diabetes
Brief Title: A Study to Compare ORMD-0801 Once Daily to ORMD-0801 Three Times Daily in Subjects With Type 1 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oramed, Ltd. (Industry)
Collaborators: Integrium (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ORA-D-017
Record Dates: First submitted 2019-10-31; First posted 2019-11-04 (Actual); Results first posted 2022-06-02 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin

STUDY DESIGN:
Intervention Model Description: This is an open-label crossover study in which all subjects will receive placebo run-in during Period 1 followed by Period 2, where subjects will be randomly assigned to either daily Treatment A (taken at Bedtime) and Treatment B (taken daily before each of three daily meals). At visit 5, the start of Period 3, subjects will stop their treatment (either A or B) and be CROSSED OVER to the other treatment (patients on treatment A during Period 2 will be crossed over to Treatment B and patients who were on Treatment B during Period 2 will be crossed over to Treatment A in Period 3).
Masking Description: Open-Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo then Treatment A then Treatment B (Experimental): Treatment administered in the following order:
  1. Period 1: Placebo (Fish Oil Capsule)
  2. Period 2: Treatment A: 24 mg ORMD-0801;(16 mg + 8 mg capsules) Once Daily (QD) at Bedtime
  3. Period 3:Treatment B: 8 mg ORMD-0801; one 8 mg capsule three times a day (TID) 45-90 minutes before meals
  Interventions: Drug: ORMD-0801 Treatment A; Drug: ORMD-0801 Treatment B; Other: Placebo
- Placebo then Treatment B then Treatment A (Experimental): Treatment administered in the following order:
  1. Period 1: Placebo (Fish Oil Capsule)
  2. Period 2:Treatment B: 8 mg ORMD-0801; one 8 mg capsule three times a day (TID) 45-90 minutes before meals
  3. Period 3: Treatment A: 24 mg ORMD-0801;(16 mg + 8 mg capsules) Once Daily (QD) at Bedtime
  Treatment B: 8 mg ORMD-0801; one 8 mg capsule three times a day (TID) 45-90 minutes before meals
  Interventions: Drug: ORMD-0801 Treatment A; Drug: ORMD-0801 Treatment B; Other: Placebo

INTERVENTIONS:
Drug: ORMD-0801 Treatment A — Treatment A: 24 mg (16 mg capsule + 8 mg capsule) Once Daily (QD) at bedtime
  Other Names: Oral Insulin
Drug: ORMD-0801 Treatment B — Treatment B: 8 mg (8 mg capsule) three times a day (TID) 45-90 minutes before meals
  Other Names: Oral Insulin
Other: Placebo — Fish oil capsule

SUMMARY:
This study is a Phase 2 randomized, crossover study comparing ORMD-0801 given QD versus TID in subjects with T1D. Subjects with T1D will have a screening visit (Visit 1) during which they will be required to review and sign the informed consent form. Medical history and demographics will be collected. Vital signs will be measured, physical exam will be performed, and blood and urine samples will be collected for hematology/chemistry/urinalysis

Placebo capsules will be given QD at bedtime during placebo run-in period 10 days prior to randomization.

DETAILED DESCRIPTION:
This study is a Phase 2 randomized, crossover study comparing ORMD-0801 given QD versus TID in subjects with T1D. Subjects with T1D will have a screening visit (Visit 1) during which they will be required to review and sign the informed consent form. Medical history and demographics will be collected. Vital signs will be measured, physical exam will be performed, and blood and urine samples will be collected for hematology/chemistry/urinalysis. Eligible subjects will be scheduled to return to the clinic in 1 week (Visit 2). Subjects fulfilling all inclusion/exclusion criteria will have a CGM placed, provided with a diary, dispensed Placebo capsules and asked to return to the clinic in 10 Days (Visit 3, Day 1) for randomization. At Visit 3, data from CGM will be downloaded and diaries will be collected. Blood samples will be collected in fasting for chemistry and HbA1c. Subjects will be randomized to receive either ORMD-0801 24 mg given once daily at bedtime, or ORMD-0801 8 mg given three times a day, 45-90 minutes before meals.

Subjects will be instructed to continue their normal diet, and to adjust their basal and bolus insulin in the normal fashion. Subjects will be instructed to return to the clinic 10 days before Visit 5 (Visit 4, Day 18). At Visit 4, compliance will be assessed, IMP and diary dispensed and the CGM will be placed. Subjects will be instructed to return to the clinic in 10 days for Visit 5 (Day 28). At Visit 5 a fasting blood sample for chemistry panel and HbA1C will be drawn and after the diary has been collected and the CGM monitor removed, they will be crossed over to the alternate treatment regimen. IMP will be dispensed, and the subject will be asked to return 10 days before Visit 7 for Visit 6 (Day 46). At Visit 6, compliance will be checked, IMP and diary will be dispensed and the CGM will be placed. Subjects will be instructed to return in 10 days for Visit 7 (Day 56). At Visit 7 the CGM will be removed, compliance checked, the diary will be collected, and a blood sample will be drawn for a chemistry panel and HbA1C. A physical examination will be performed, and the subject will exit the study. Subjects will be provided with diaries at Visits 2, 4 and 6, and will be asked to capture the amount of basal and bolus exogenous insulin administered each day and calculate their carbohydrate count for all meals and snacks over the 10-day CGM monitoring period. Diaries will be collected at Visits 3, 5 and 7.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged 18 and older.
* Body mass index (BMI) of 19-30 kg/m2 at Screening and stable weight, with no more than 5 kg gain or loss in the 3 months prior to Screening.
* T1D subjects must have:

  1. A documented history of type 1 diabetes for at least 6 months
  2. Should be on an MDI regimen
  3. C peptide levels of ˂ 0.7 ng/mL
  4. HbA1C ≥ 6.5% to ≤10%
* Females of childbearing potential must have a negative serum pregnancy test result at Screening.
* Females who are not of childbearing potential are defined as:

  1. post-menopausal (defined as at least 12 months with no menses in women ≥45 years of age) or
  2. has had a hysterectomy and/or bilateral oophorectomy, or had bilateral tubal ligation or occlusion at least 6 weeks prior to Screening
* Subjects who are of childbearing potential must:

  a. agree to remain abstinent from heterosexual activity† or agree to use (or have their partner use) acceptable contraception to prevent pregnancy within the projected duration of the trial and for 14 days after the last dose of blinded investigational product. Two methods of contraception will be used to avoid pregnancy. Acceptable combinations of methods include: i. Use of one of the following double-barrier methods: diaphragm with spermicide and a condom; cervical cap and a condom; or a contraceptive sponge and condom ii. Use of hormonal contraception (any registered and marketed contraceptive agent that contains an estrogen and/or a progestational agent [including oral, subcutaneous, intrauterine and intramuscular agents, and cutaneous patch]) with one of the following: diaphragm with spermicide; cervical cap; contraceptive sponge; condom; vasectomy; or IUD. iii. Use of an IUD with one of the following: condom; diaphragm with spermicide; contraceptive sponge; vasectomy; or hormonal contraception (see above).

iv. Vasectomy with one of the following: diaphragm with spermicide; cervical cap; contraceptive sponge; condom; IUD; or hormonal contraception (see above).

†Abstinence can be used as the sole method of contraception if it is in line with the subject's preferred and usual lifestyle and if considered acceptable by local regulatory agencies and ethics committees. Periodic abstinence (e.g., calendar, ovulation, sympto-thermal, post-ovulation methods, etc.) and withdrawal are not acceptable methods of contraception.

Exclusion Criteria:

* Clinical diagnosis of type 2 diabetes;
* Evidence of unawareness of hypoglycemia unawareness, a documented plasma glucose ≤50 mg/dL in the absence of symptoms of hypoglycemia at Screening.
* FPG >300 mg/dL at Screening; a single repeat test is allowable.
* Use of the following medications:

  1. Administration of thyroid preparations or thyroxine (except in subjects on stable replacement therapy) within 6 weeks prior to Screening.
  2. Administration of systemic long-acting corticosteroids within two months or prolonged use (more than one week) of other systemic corticosteroids or inhaled corticosteroids (if daily dosage is > 1,000 μg equivalent beclomethasone) within 30 days prior to Screening. Intra-articular and/or topical corticosteroids are not considered systemic.
* Laboratory abnormalities at Screening including:

  1. Abnormal serum thyrotropin (TSH) levels below the lower limit of normal or >1.5X the upper limit of normal
  2. Elevated liver enzymes (alanine transaminase (ALT), alanine aminotransferase (AST), alkaline phosphatase) >2X the upper limit of normal.
  3. Very high triglyceride levels (>600 mg/dL); a single repeat test is allowable.
  4. Any relevant abnormality that would interfere with the efficacy or the safety assessments during study treatment administration.
* Subject has a Screening systolic blood pressure ≥165 mmHg or diastolic blood pressure ≥100 mmHg. Subjects will be allowed to take a BP rescue medication.
* Any clinically significant ECG abnormality at Screening or cardiovascular disease. Clinically significant cardiovascular disease will include:

  a. History of stroke, transient ischemic attack, or myocardial infarction within 6 months prior to Screening,
* History of or currently have New York Heart Associate Class II-IV heart failure prior to Screening.
* Presence of any clinically significant endocrine disease according to the Investigator (euthyroid subjects on replacement therapy will be included if the dosage of thyroxine is stable for at least six weeks prior to Screening).
* Presence of any clinically significant condition (in the opinion of the Investigator) that might interfere with the evaluation of study medication, such as significant renal, hepatic, gastrointestinal (GI), cardiovascular (CV), immune disease, blood dyscrasias or any disorders causing hemolysis or unstable red blood cells, or clinically important hematological disorders (i.e. aplastic anemia, myeloproliferative or myelodysplastic syndromes, thrombocytopenia) at Screening.
* History of gastrointestinal disorders (e.g. hypochlorhydria) with the potential to interfere with drug absorption.
* Presence or history of cancer within the past 5 years of Screening, with the exception of adequately-treated localized basal cell skin cancer or in situ uterine cervical cancer.

  1. A subject with a history of malignancy >5 years prior to Screening should have no evidence of residual or recurrent disease.
  2. A subject with a history of melanoma, leukemia, lymphoma, or renal carcinoma is excluded.
* Positive history of active liver disease (other than non-alcoholic hepatic steatosis), including chronic hepatitis B or C, primary biliary cirrhosis, or active symptomatic gallbladder disease.
* Positive history of HIV.
* Known allergy to soy.
* Subject is on a weight loss program and is not in the maintenance phase, or subject has started weight loss medication (e.g., orlistat or liraglutide), within 8 weeks prior to Screening. Subjects who have had bariatric surgery are also excluded.
* S ubject is pregnant or breast-feeding.
* Subject is a user of recreational or illicit drugs or has had a recent history (within 1 year of Screening) of drug or alcohol abuse or dependence. (Note: Alcohol abuse includes heavy alcohol intake as defined by >3 drinks per day or >14 drinks per week, or binge drinking) at Screening.
* At the Principal Investigator's discretion, any condition or other factor that is deemed unsuitable for subject enrollment into the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-10-17 (Actual); Primary Completion 2020-02-06 (Actual); Study Completion 2020-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Kidron, PhD, Study Director — Oramed Pharmaceuticals, Inc.
Locations (1):
- Orange County Research Center, Tustin, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a crossover study with one crossover point.
  There are three periods in this study:
  Period 1: all patients consented receive placebo (run-in period). Period 2: all patients are randomized to receive either Treatment A or Treatment B.
  Period 3: Crossover point. Patients receiving Treatment A in period 2 now receive Treatment B in period 3, and patients receiving Treatment B in period 2 now receive Treatment A in period 3.
Groups:
- Placebo Followed by Treatment A Followed by Treatment B: Treatment administered in the following order:
  1. Placebo Fish oil capsule
  2. Treatment A is 24 mg (16 mg + 8 mg capsules) Once Daily (QD) at Bedtime of ORMD-0801 ORMD-0801: Oral Insulin Capsules
  3. Treatment B is 8 mg (8 mg capsule) three times a day (TID) 45-90 minutes before meals ORMD-0801: Oral Insulin Capsules
- Placebo Followed by Treatment B Followed by Treatment A: Treatment administered in the following order:
  1. Placebo Fish oil capsule
  2. Treatment B is 8 mg (8 mg capsule) three times a day (TID) 45-90 minutes before meals ORMD-0801: Oral Insulin Capsules
  3. Treatment A is 24 mg (16 mg + 8 mg capsules) Once Daily (QD) at Bedtime of ORMD-0801 ORMD-0801: Oral Insulin Capsules
Period: Period 1- Placebo run-in (All Patients)
Arm/Group | Placebo Followed by Treatment A Followed by Treatment B | Placebo Followed by Treatment B Followed by Treatment A
Started | 14 | 16
Completed | 14 | 16
Not Completed | 0 | 0
Period: Period 2- Either Treatment A or B
Arm/Group | Placebo Followed by Treatment A Followed by Treatment B | Placebo Followed by Treatment B Followed by Treatment A
Started | 14 | 16
Completed | 14 | 16
Not Completed | 0 | 0
Period: Period 3 Crossover-Treatment B or A
Arm/Group | Placebo Followed by Treatment A Followed by Treatment B | Placebo Followed by Treatment B Followed by Treatment A
Started | 14 | 16
Completed | 12 | 15
Not Completed | 2 | 1
Not completed — Adverse Event | 2 | 0
Not completed — Patient non-compliance | 0 | 1

BASELINE CHARACTERISTICS:
Population: All patients are first administered a placebo, or is the standard of care.
Groups:
- Placebo Followed by Treatment A Followed by Treatment B: Treatment administerd in the following order:
  1. Placebo, standard of care Fish oil capsules
  2. Treatment A is 24 mg (16 mg + 8 mg capsules) Once Daily (QD) at Bedtime of ORMD-0801 ORMD-0801: Oral Insulin Capsules
  3. Treatment B is 8 mg (8 mg capsule) three times a day (TID) 45-90 minutes before meals ORMD-0801: Oral Insulin Capsules
- Placebo Followed by Treatment B Followed by Treatment A: Treatment administerd in the following order:
  1. Placebo, standard of care Fish oil capsules
  2. Treatment B is 8 mg (8 mg capsule) three times a day (TID) 45-90 minutes before meals ORMD-0801: Oral Insulin Capsules
  3. Treatment A is 24 mg (16 mg + 8 mg capsules) Once Daily (QD) at Bedtime of ORMD-0801 ORMD-0801: Oral Insulin Capsules
- Total: Total of all reporting groups
Arm/Group | Placebo Followed by Treatment A Followed by Treatment B | Placebo Followed by Treatment B Followed by Treatment A | Total
Number analyzed (Participants) | 14 | 16 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: This is a crossover study. All patients were administered placebo at baseline.
  years | 43.79285714 (12.67793142) | 42.88125 (16.04131614) | 43.30667 (12.22325)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 7 | 8 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 13 | 15 | 28
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 14 | 14 | 28
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Pre-dose Hb1Ac(%) [Mean (Standard Deviation); unit: percent] — Hb1Ac is a measurement from a blood sample of the glycated form of hemoglobin to obtain the two to three-month average of blood sugar. the inclusion criterion for Hb1Ac is 6.5% ≤ HbA1c ≤10%
  percent | 7.735714286 (0.734435569) | 7.6125 (0.848429922) | 7.67 (0.786)

OUTCOME MEASURES:

1. Primary Outcome: Average Exogenous Basal Insulin Compared to Baseline (Placebo)
Description: The least squares means difference of basal exogenous insulin between treatment A and placebo and treatment B and placebo, utilized over the final ten (10) days of each treatment period
Time Frame: Combined Final ten days of each treatment period. Period1 (days -8 to 1)Period 2 (days 19 to 28) ,and Period 3 (days 47 to 56)
Population: Information collected at the day 28 visits (Day 28 and Day 56) will be analyzed using an Analysis of Covariance model with subject as a random effect.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Groups:
- Baseline: Placebo (Fish-Oil Capsule)
- Treatment A: Treatment A is 24 mg (16 mg + 8 mg capsules) Once Daily (QD) at Bedtime of ORMD-0801
  ORMD-0801: Oral Insulin Capsules
- Treatment B: Treatment B is 8 mg (8 mg capsule) three times a day (TID) 45-90 minutes before meals
  ORMD-0801: Oral Insulin Capsules
Arm/Group | Baseline | Treatment A | Treatment B
Number analyzed (Participants) | 30 | 27 | 27
mg/dL
  Least Squares Mean Baseline, Treatment A, Treatment B | 27.28 (2.489) | 25.84 (2.486) | 27.32 (2.492)
  Least Squares Mean Difference Treatment A minus Baseline or Treatment B minus Baseline | NA (NA) — Calculation not applicable to this Arm/Group | -1.43 (0.381) | 0.04 (0.421)
Statistical Analysis 1: Comparison: Baseline vs Treatment A vs Treatment B; Information collected in the daily diaries or via the Continuous Glucose Monitor (CGM) on the final 10 days of treatment will be analyzed using a Repeated Measures Analysis of Covariance with subject as a random effect with each of the 10 days being a single measurement. When analyzing the exogenous insulin variables, the CGM parameters (mean 24 hour glucose value and 24 hour time within 70-180 mg/dL range) and the patient reported carbohydrate intake will be included as covariates; Test type: Other — Treatment least squares means and change from baseline estimates will be derived using this linear model; p < 0.9223, ANCOVA; Least mean squares

2. Primary Outcome: Average Exogenous Bolus Insulin Compared to Baseline (Placebo)
Description: The amount of exogenous bolus insulin utilized over the final ten (10) days of each treatment period measured in mg/dL
Time Frame: Combined Final ten days of treatment per treatment period (Days -8 to 1, Days 19 to 28, and Days 47 to 56)
Population: Safety Population
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Baseline | Treatment A | Treatment B
Number analyzed (Participants) | 30 | 27 | 27
mg/dL
  Least Squares Means Baseline, Treatment A, Treatment B | 20.63 (2.033) | 20.77 (2.045) | 20.54 (2.049)
  Least Squares Means Difference Treatment A minus Baseline, Treatmen B minus Baseline | NA (NA) — Calculation not applicable to this Arm/Group. | 0.14 (0.634) | -0.09 (0.645)
Statistical Analysis 1: Comparison: Baseline vs Treatment A vs Treatment B; [analysis description as in outcome 1, analysis 1]; Test type: Other — Treatment least squares means and change from baseline estimates will be derived using this linear model; p < 0.8871, ANCOVA

3. Primary Outcome: Average Exogenous Total Insulin Compared to Baseline
Description: The Least Squares Mean Difeerence ( (mg/dL) of total exogenous insulin (the sum of basal + bolus exogenous insulin) over the final ten (10) days of treatment.
Time Frame: Combined Final ten days of treatment , day -8 to 1 (Period 1) Days 19 to 28 (Period 2), Days 47 to 56 (Period 3)
Population: Safety Population The number of participants anylized is based on the the number of participants that completed at least 80% of the Continuous Glucose Montioring measurements. Participants that did not meet this criterion are not inclued in this analysis.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Baseline | Treatment A | Treatment B
Number analyzed (Participants) | 29 | 27 | 27
mg/dL
  Least Squares Mean | 47.92 (3.395) | 46.64 (3.397) | 47.88 (3.406)
  Least Squares Mean Difference Treatment A minus Baseline and Treatment B minus Baseline | NA (NA) — Calculation not applicable to this Arm/Group. | -0.127 (0.758) | -0.04 (0.798)
Statistical Analysis 1: Comparison: Baseline vs Treatment A vs Treatment B; [analysis description as in outcome 1, analysis 1]; Test type: Other — Treatment least squares means and change from baseline estimates will be derived using this linear model; p < 0.9641, ANCOVA

4. Secondary Outcome: Daytime Average Mean Glucose Compared to Baseline
Description: Least Squares Mean Difference from Baseline of Daytime Average Mean Glucose over the final ten (10) days of each treatment and each treatment period as measured by CGM.
Time Frame: Combined Study days -8 to 1 (Period 1) Days 19 to 28 (Period 2), and days 47 to 56 (Period 3)
Population: Safety Population. The number of participants anylized is based on the the number of participants that completed at least 80% of the Continuous Glucose Montioring measurements. Participants that did not meet this criterion are not inclued in this analysis.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Baseline | Treatment A | Treatment B
Number analyzed (Participants) | 30 | 26 | 26
mg/dL
  Least Sqaures Mean Baseline, Treatment A, Treatment B | 168.72 (5.825) | 174.84 (5.957) | 169.75 (5.930)
  Least Squares Mean Difference between each treatment and placebo | NA (NA) — Calculation not applicable to this Arm/Group. | 6.12 (3.966) | 1.02 (3.889)
Statistical Analysis 1: Comparison: Baseline vs Treatment A vs Treatment B; [analysis description as in outcome 1, analysis 1]; Test type: Other — Treatment least squares means and change from baseline estimates will be derived using this linear model; p < 0.7922, ANCOVA

5. Secondary Outcome: Daytime Glucose Coefficient of Variation Compared to Baseline
Description: Least Squares Mean Continuous Glucose Monitor (CGM) Glucose Coefficient of Variation measured over daytime hours, compared to Baseline
Time Frame: Study Days -8 to 1 (Period 1), Days 19-28 (Period 2), and Days 47-56 (Period 3)
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: percent (%)
Arm/Group | Baseline | Treatment A | Treatment B
Number analyzed (Participants) | 30 | 26 | 26
percent (%)
  Least Squares Mean | 45.287 (2.3191) | 46.550 (2.3073) | 44.996 (2.2847)
  Least Squares Mean Differece between each treatment and placebo. | NA (NA) — Calculation not applicable to this Arm/Group. | 1.64 (1.949) | -0.291 (1.9064)
Statistical Analysis 1: Comparison: Baseline vs Treatment A vs Treatment B; [analysis description as in outcome 1, analysis 1]; Test type: Other — Treatment least squares means and change from baseline estimates will be derived using this linear model; p < 0.9898, ANCOVA

6. Secondary Outcome: Daytime Low Blood Glucose Index (LBGI) Compared to Baseline
Description: Least Squares Mean Daytime Low Blood Glucose Index (LBGI) measured over the last ten (10) days of the treatment period, compared to Baseline LBGI is a clinical scale that indicates the probability for hypoglycemia. Blood Glucose Variability is an important measure because it provides additional clarification for HbA1c value.
  The risk of hypglycemic events and the LBGI scale is defined as follows:
  Minimal Risk ( LBGI < 1.1) Low Risk ( 1.1 < LBGI < 2.5) Moderate Risk (2.5 < LBGI < 5), HIgh Risk ( LBGI > 5)
Time Frame: Combined Study Days -8 to 1 (Period 1), Days 19-28 (Period 2), and Days 47-56 (Period 3)
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Baseline | Treatment A | Treatment B
Number analyzed (Participants) | 30 | 26 | 26
units on a scale
  Least Squares Mean Daytime Low Blood Glucose Index (LBGI) for Baseline, | 1.65 (0.284) | 1.53 (0.282) | 1.65 (0.288)
  Least Squares Mean Difference between Treatment A and Placebo, Treatment B and Placebo. | NA (NA) — Calculation not applicable to this Arm/Group. | -0.12 (0.294) | 0.00 (0.297)
Statistical Analysis 1: Comparison: Baseline vs Treatment A vs Treatment B; [analysis description as in outcome 1, analysis 1]; Test type: Other — Treatment least squares means and change from baseline estimates will be derived using this linear model; p < 0.5165, ANCOVA

ADVERSE EVENTS:
Time Frame: Sixty-six (66) days
Groups:
- Placebo: Placebo - Fish Oil
- Treatment A ORMD-0801: Treatment A is 24 mg (16 mg + 8 mg capsules) Once Daily (QD) at Bedtime of ORMD-0801
  ORMD-0801 Treatment A: Treatment A: 24 mg (16 mg capsule + 8 mg capsule) Once Daily (QD) at bedtime
- Treatment B ORMD-0801: Treatment B is 8 mg (8 mg capsule) three times a day (TID) 45-90 minutes before meals
  ORMD-0801 Treatment B: Treatment B: 8 mg (8 mg capsule) three times a day (TID) 45-90 minutes before meals
Arm/Group | Placebo | Treatment A ORMD-0801 | Treatment B ORMD-0801
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 9/30 | 6/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=30) | Treatment A ORMD-0801 (N=30) | Treatment B ORMD-0801 (N=30)
Nasopharangitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — mild
OTITIS EXTERNA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — mild
Sinusitis (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) — mild
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) — mild
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) — mild
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) — mild
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) — moderate
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) — severe
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) — mild
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — mild

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2019-08-29): https://cdn.clinicaltrials.gov/large-docs/07/NCT04150107/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-09): https://cdn.clinicaltrials.gov/large-docs/07/NCT04150107/SAP_001.pdf